CLINICAL TRIAL: NCT01620931
Title: A Single-Center, Randomized, Observer-Blinded, Placebo-Controlled, Single-Ascending-Dose (SAD) Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO5469754, a Humanized Monoclonal Antibody, Following Intravenous or Subcutaneous Administration in Healthy Adults
Brief Title: A Single-Ascending-Dose Study of RO5469754 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NP27885
Record Dates: First submitted 2012-06-06; First posted 2012-06-15 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RO5469754 (Experimental)
  Interventions: Drug: RO5469754

INTERVENTIONS:
Drug: Placebo — Single doses, iv or sc
  Arms: Placebo
Drug: RO5469754 — Single ascending doses, iv or sc
  Arms: RO5469754

SUMMARY:
This randomized, observer-blinded, placebo-controlled study will assess the safety, tolerability, pharmacokinetics and pharmacodynamics of RO5469754 in healthy volunteers. Subjects will be randomized in cohorts to receive single ascending intravenous or subcutaneous doses of RO5469754 or placebo. In-clinic period will be from Day -1 to Day 4, with a safety follow-up of 15 weeks after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers, 18 to 64 years of age, inclusive
* Body mass index (BMI) 18 to 32 kg/m2
* Women of child-bearing potential and their partners must be willing to use two highly effective forms of contraception, one of which must be a barrier method, for the entire duration of the study (through study discharge) or for up to five half-lives after the last dose
* Male subjects with female partners of child-bearing potential must be willing to use a condom during sexual activity for the duration of the study (through study discharge) or for up to five half-lives after the last dose

Exclusion Criteria:

* Pregnant or lactating women
* Positive test for drugs of abuse (including ethanol) as per local standards
* Willing to comply with a non-smoking policy during the in-clinic part of the study (Day -1 until discharge on Day 4)
* Positive for hepatitis B, hepatitis C or HIV infection
* History or presence of clinically significant disease or condition
* Participation in an investigational drug or device study within 60 days prior to dosing
* Current (or previous history of) exposure to therapeutic or investigational monoclonal antibody or chimeric biomolecule
* Any confirmed clinically significant previous allergic drug reaction, or history of anaphylaxis

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-11-07 (Actual); Primary Completion 2012-09-03 (Actual); Study Completion 2012-09-03 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 1 year

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve (AUC) | Pre-dose and up to 72/120 hours post-dose, and at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Groningen, Netherlands